CLINICAL TRIAL: NCT01434121
Title: Ascorbic Acid (Vitamin C) Infusion in Human Sepsis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM12903
Record Dates: First submitted 2011-08-09; First posted 2011-09-14 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Sepsis; Septic Shock; Hypotension; Acute Lung Injury
MeSH Terms: conditions — Sepsis; Shock, Septic; Hypotension; Acute Lung Injury | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Dose Ascorbic Acid (Active Comparator): Subject receives a high dose of infused Vitamin C
  Interventions: Drug: Ascorbic Acid
- Low Dose Ascorbic Acid (Active Comparator): Subject receives a low dose of infused Vitamin C
  Interventions: Drug: Ascorbic Acid
- Placebo (Placebo Comparator): Subject receives an infusion of saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ascorbic Acid — The infusion of either a high dose of ascorbic acid, low dose ascorbic acid, or placebo
  Other Names: Vitamin C
  Arms: High Dose Ascorbic Acid; Low Dose Ascorbic Acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
The major goal of this project is to determine whether intravenously infused ascorbic acid is safe for use as a viable therapeutic strategy in adult humans with sepsis.

DETAILED DESCRIPTION:
Evolving data from experimental animals strongly suggests that ascorbic acid potently interrupts multiple biological processes which lead to organ injury following onset of sepsis. Data presented below suggests that ascorbic acid potently attenuates lung injury produced by septic insults. Sepsis and septic shock secondary to bacterial and fungal blood stream infections are a leading cause of death in critically ill patients. At present, 28 day mortality in septic patients averages 40% in the best of ICUs. In sepsis, disseminated intravascular coagulation produces widespread systemic microvascular thrombosis that leads to multiple organ injury (i.e., lung, liver, kidney, intestinal, cardiovascular). Despite aggressive intravascular volume resuscitation and vasopressor support, appropriate antibiotic administration, and expert critical care management, mortality remains high. Only a single agent has been approved to disrupt progressive sepsis-associated microvascular thrombosis (activated protein C, [Drodrecogin Alpha, brand name: Xigris, Lilly]). No other non-antibiotic pharmaceutical agent is currently approved for use in sepsis. Activated protein C (APC) continuous infusion protocol spans a 96 hour period. APC infusion produces significant anticoagulation, and therefore the major risk from its use is hemorrhage. Thus, recent surgery, especially neurosurgical procedures, is a major contraindication to APC use. Finally, cost stands as an important issue for APC use. A 96 hour APC infusion in a 70 kg patient at VCUHS costs the patient over $33,000 (source VCUHS Pharmacy Services). Use of APC in sepsis remains controversial and has failed to achieve widespread acceptance. The goal of the current study is to determine the safety of ascorbic acid infusion in septic humans.

ELIGIBILITY:
Inclusion Criteria:

1. systemic inflammatory response: fever (38°C or greater) or hypothermia (36°C or lower), tachypnea (20 breaths/min) or need for mechanical ventilation for an acute process, tachycardia (rate 90/min or more), white blood cell count ≥ 12,000 cells/mm3 or ≤ 4,000 cells/mm3 or more than 10% band forms.
2. Presumed or Known Site of Infection: Purulent sputum, chest radiograph with new infiltrate, spillage of bowel contents, radiographic or physical examination evidence of an infected collection, white blood cells in a normally sterile body fluid, positive blood culture, evidence of infected mechanical hardware by physical, radiographic, or ultrasonographic evidence.
3. Evidence of Dysfunction of One or More End Organs: cardiovascular dysfunction: mean arterial pressure 60 mm Hg or less, the need for vasopressors to maintain this pressure in the presence of adequate intravascular volume (central venous pressure 12 mmHg); respiratory failure: (arterial PO2-to-FiO2 ratio of less than 250 or less than 200 in the presence of pneumonia; renal dysfunction: Urine output ≤ 0.5 ml/kg/hr for 2 hours in the presence of adequate intravascular volume or doubling of the serum creatinine; hematologic dysfunction: thrombocytopenia ≤ 80,000 platelets/mm3 or 50% decrease from baseline during the acute illness; Unexplained metabolic acidosis: arterial pH ≤ 7.3 and a plasma lactate level higher than 2.5. Hepatic Dysfunction: Acute Serum transaminase elevation greater than five times normal.
4. Informed Consent: Ability to obtain informed consent within 48 hours.

Exclusion Criteria:

1. Demographic Characteristics: Children (age < 18 years), pregnant women, prisoners, and other wards of the state are excluded from participation in this study.
2. Informed Consent: Inability to obtain informed consent within 48 hours.
3. Cognitive Impairment: In the absence of family or next of kin, if the investigators feel the patient is cognitively impaired, and unable to provide informed consent, the patient will not be accessed to the study.
4. Non-English Speaking Patients: Patients who are non english speaking will not be accessed to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alpha Fowler, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Ascorbic Acid: Subject receives a high dose of infused Vitamin C
  Ascorbic Acid vs. Placebo: The infusion of either a high dose of ascorbic acid, low dose ascorbic acid, or placebo
- Low Dose Ascorbic Acid: Subject receives a low dose of infused Vitamin C
  Ascorbic Acid vs. Placebo: The infusion of either a high dose of ascorbic acid, low dose ascorbic acid, or placebo
- Placebo: Subject receives an infusion of saline
  Ascorbic Acid vs. Placebo: The infusion of either a high dose of ascorbic acid, low dose ascorbic acid, or placebo
Period: Overall Study
Arm/Group | High Dose Ascorbic Acid | Low Dose Ascorbic Acid | Placebo
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Ascorbic Acid | Low Dose Ascorbic Acid | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 6 | 19
  >=65 years | 2 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 11
  Male | 4 | 5 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 3 | 10
  White | 5 | 4 | 5 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 2 | 11
  Unknown or Not Reported | 4 | 3 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced Ascorbic Acid Infusion Related Arterial Hypotension, Vomiting, or Tachycardia in Septic Patients
Description: There were no instances of arterial hypotension, vomiting, or tachycardia within the study population related to the study drug
Time Frame: during time of infusion- 96 hours from time of enrollment
Measure: Number; unit: participants
Arm/Group | High Dose Ascorbic Acid | Low Dose Ascorbic Acid | Placebo
Number analyzed (Participants) | 8 | 8 | 8
participants | 0 | 0 | 0

2. Secondary Outcome: Intensive Care Unit Length of Stay
Time Frame: subject will be followed until discharged from the ICU, has deceased, or study duration has reached 28 days from time of enrollment, whichever is first
Population: Limited data were collected for this assessment due to study termination. These data are no longer available and the study team does not have IRB approval to retroactively analyze the results
Groups:
- Placebo: Subject receives an infusion of saline
  Placebo
Arm/Group | High Dose Ascorbic Acid | Low Dose Ascorbic Acid | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Duration of Mechanical Ventilation
Time Frame: subject will be followed until mechanical ventilation has been discontinued, the subject has deceased, or study duration has reached 28 days from time of enrollment, whichever is first
Population: as for outcome 2
Arm/Group | High Dose Ascorbic Acid | Low Dose Ascorbic Acid | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Ventilator-free Days
Time Frame: subject will be followed until discharged from the hospital, has deceased, or study duration has reached 28 days from time of enrollment, whichever is first
Population: as for outcome 2
Arm/Group | High Dose Ascorbic Acid | Low Dose Ascorbic Acid | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Length of Time on Vasopressor Medication
Time Frame: during time of infusion - 96 hours from time of enrollment
Population: as for outcome 2
Arm/Group | High Dose Ascorbic Acid | Low Dose Ascorbic Acid | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Multiple Organ Dysfunction Score
Time Frame: during time of infusion - 96 hours from time of enrollment
Population: as for outcome 2
Arm/Group | High Dose Ascorbic Acid | Low Dose Ascorbic Acid | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Plasma Cytokine/Chemokine Levels
Time Frame: during time of infusions - 96 hours from time of enrollment
Population: as for outcome 2
Arm/Group | High Dose Ascorbic Acid | Low Dose Ascorbic Acid | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 96 hours
Arm/Group | High Dose Ascorbic Acid | Low Dose Ascorbic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes